CLINICAL TRIAL: NCT01353248
Title: A Phase 2 Randomized, Open-Label Study of GS-5885 Administered Concomitantly With GS-9451, Tegobuvir and Ribavirin (RBV) to Treatment-Naive Subjects With Chronic Genotype 1 HCV Infection
Brief Title: GS 5885 Administered Concomitantly With GS-9451, Tegobuvir and Ribavirin (RBV) in Chronic Genotype 1 Hepatitis C Virus (HCV) Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-248-0120
Record Dates: First submitted 2011-04-22; First posted 2011-05-13 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-11

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C; HCV; Rapid Virologic Response; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy; HCV RNA; Polymerase inhibitor; Protease inhibitor; Treatment naïve; GS-5885; GS-9451; Tegobuvir
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — ledipasvir; tegobuvir; GS-9451; Ribavirin

ARMS (2):
- Arm 1 (Active Comparator): GS-5885, GS-9451 and Tegobuvir in combination with ribavirin (Copegus®) for 24 weeks.
  Interventions: Drug: GS-5885; Drug: Tegobuvir; Drug: GS-9451; Drug: ribavirin tablet
- Arm 2 (Active Comparator): GS-5885, GS-9451 and Tegobuvir in combination with ribavirin (Copegus®) for 12 or 24 weeks.
  Interventions: Drug: Tegobuvir; Drug: GS-9451; Drug: ribavirin tablet; Drug: GS-5885

INTERVENTIONS:
Drug: GS-5885 — tablet, 30 mg QD
  Arms: Arm 1
Drug: Tegobuvir — capsule, 30 mg BID
Drug: GS-9451 — tablet, 200 mg QD
Drug: ribavirin tablet — (weight based: 1000 mg/day <75 kg; 1200 mg/day ≥ 75 kg) divided twice daily (BID)
Drug: GS-5885 — tablet, 90 mg QD
  Arms: Arm 2

SUMMARY:
The purpose of this phase 2 study is to determine whether 30 mg or 90 mg of GS-5885 when given with GS-9451, Tegobuvir and Ribavirin (RBV) for 12 or 24 weeks is effective, safe and tolerable in the treatment of Chronic Genotype 1 HCV Infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects 18 to 70 years of age
* Chronic HCV infection for at least 6 months prior to Baseline (Day 1)
* Liver biopsy results (performed no more than 2 years prior to Screening) indicating the absence of cirrhosis
* Monoinfection with HCV genotype 1a or 1b
* HCV treatment-naïve
* Body mass index (BMI) between 18 and 36 kg/m2
* Creatinine clearance ≥ 50 mL/min
* Subject agrees to use highly effective contraception methods if female of childbearing potential or sexually active male.
* Screening laboratory values within defined thresholds

Exclusion Criteria:

* Autoimmune disease
* Decompensated liver disease or cirrhosis
* Poorly controlled diabetes mellitus
* Severe psychiatric illness
* Severe chronic obstructive pulmonary disease (COPD)
* Serological evidence of co-infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or another HCV genotype
* Suspicion of hepatocellular carcinoma or other malignancy (with exception of certain skin cancers)
* History of hemoglobinopathy
* Known retinal disease
* Subjects who are immunosuppressed
* Subjects with known, current use of amphetamines, cocaine, opiates (i.e., morphine, heroin), methadone, or ongoing alcohol abuse
* Subjects must have no history of clinically significant cardiac disease, including a family history of Long QT syndrome, and no relevant electrocardiogram (ECG) abnormalities at screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2011-05; Primary Completion 2012-10 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response (SVR) | 24 weeks of off-treatment follow-up

SECONDARY OUTCOMES:
Safety and tolerability | through 24 weeks of off-treatment follow-up
  To evaluate the safety and tolerability of 30 mg or 90 mg GS-5885 when given with GS-9451, Tegobuvir and RBV for 12 or 24 weeks. Safety endpoints will be analyzed by the number and percent of subjects with events or abnormalities for categorical values or 8-number summary (n, mean, standard deviation, median, Q1, Q3, minimum, maximum) for continuous data by treatment group.
HCV RNA < Lower Limit Of Quantification | Weeks 1, 2, 4, 12 and 24
  To evaluate the antiviral efficacy at Weeks 1, 2, 4, 12 and 24, as measured by the rates of HCV RNA < LLoQ and viral breakthrough and relapse.
Rescue Therapy Substudy SVR | 24 Weeks
  To evaluate the antiviral efficacy (as defined by SVR) of the addition of pegylated interferon (PEG) for 24 weeks to GS-5885, GS-9451, tegobuvir and RBV in subjects who experience viral breakthrough on treatment.
Emergence of viral resistance | 12 or 24 weeks
  To evaluate the emergence of viral resistance during treatment with GS-9451, Tegobuvir and RBV when given with 30 mg or 90 mg GS-5885 for 12 or 24 weeks.
Viral dynamics of GS-5885, GS-9451 and Tegobuvir when administered in combination with RBV | Through Week 2 of therapy
  HCV RNA levels, pharmacokinetics and viral sequencing
Pharmacokinetics of GS-5885, GS-9451 and Tegobuvir when administered in combination with RBV | Through Week 2 of therapy
  Pharmacokinetics (Cmax, Tmax, Clast, Tlast, Ctau, λz, AUCtau, and T½) will be listed
  and summarized for GS-5885, GS-9451 and Tegobuvir using descriptive statistics (e.g.,
  sample size, arithmetic mean, geometric mean, % coefficient of variation, standard deviation,
  median, minimum, and maximum). Plasma concentrations of the study drug over time will be
  summarized using descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Benedetta Massetto, MD, PhD, Study Director — Gilead Sciences
Locations (43):
- United States (42):
  - Birmingham Gastroenterology Associates, P.C., Birmingham, Alabama
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Advanced Clinical Research Institute, Anaheim, California
  - Southern California Liver Centers, Coronado, California
  - UCSF Fresno Medical Education Program (MEP), Fresno, California
  - Stanford University School of Medicine, Palo Alto, California
  - University of California San Diego, San Diego, California
  - Kaiser Permanente, San Diego, California
  - UCSF, San Francisco, California
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Bach and Godofsky Infectious Diseases, Bradenton, Florida
  - University of Florida - Gainesville, Gainesville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Gastrointestinal Specialists of Georgia PC, Marietta, Georgia
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Private Practice, Opelousas, Louisiana
  - Johns Hopkins University, Lutherville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Gastrointestinal Associates, PA, Jackson, Mississippi
  - University of New Mexico, Albuquerque, New Mexico
  - Mount Sinai Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Options Health Research, LLC, Tulsa, Oklahoma
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Gastro One, Germantown, Tennessee
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - Columbia Medical Group, The Frist Clinic, Nashville, Tennessee
  - Nashville Gastrointestinal Specialists, Inc, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Research Specialists of Texas, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Lifetree Clinical Research, LC, Salt Lake City, Utah
  - Inova Fairfax Hospital - Center for Liver Diseases, Falls Church, Virginia
  - Liver Institute of Virginia, Bon Secours Health System, Newport News, Virginia
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico